CLINICAL TRIAL: NCT05805267
Title: To Evaluate the Correlation Between the Results of Specific Gene Testing and the Efficacy of Targeted Therapy in Patients With Non-small Cell Lung Cancer (NSCLC)
Brief Title: To Evaluate the Correlation Between the Results of Specific Gene Testing and the Efficacy of Targeted Therapy in Patients With NSCLC
Status: Completed | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Other Study IDs: CONFIDENCE II
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue sample and plasma DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluated the correlation between the qualitative test results of Xiamen Aide the gene test specified by the test reagent and the efficacy of relevant targeted drugs in patients with non-small cell lung cancery, and the research data is used to support the registration and marketing of the assessment reagent

ELIGIBILITY:
Inclusion Criteria:

* 1)≥18;
* 2) advanced non-small cell lung cancer confirmed by histopathology;
* 3) Patients with NSCLC who have previously or are taking gefitinib (first-line therapy) or osimertinib (post-TKI resistance) or crizotinib monotherapy, and the response to treatment can be assessed;
* 4) Have sufficient FFPE tissue samples within 5 years: 5 large specimens/case; There were 10 puncture specimens/case

Exclusion Criteria:

* 1) Combination therapy with chemotherapy/radiotherapy/other targeted drugs/immunotherapy drugs;
* 2)Maintenance therapy if the disease does not progress after treatment with other antitumor methods

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer who have previously received or are taking gefitinib (first-line therapy) or osimertinib (post-TKI resistance) or crizotinib monotherapy
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
PFS | 2 year
  Defined as the time from the beginning of treatment to the first imaging disease progression or death (whichever occurs first)

SECONDARY OUTCOMES:
ORR | 2 years
  Defined as the proportion of subjects in complete remission (CR) and partial remission (PR) to the total subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China